CLINICAL TRIAL: NCT02891486
Title: Analysis of the Incidence of Post-Operative Wound Infections After Spine Surgery - a Prospective Study
Brief Title: Analysis of the Incidence of Post-Operative Wound Infections After Spine Surgery
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Allan D. Levi, MD, PhD, Professor and Chairman of Neurological Surgery, University of Miami
Other Study IDs: 20110185
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Infection
Keywords: spinal surgery, surgical site infection
MeSH Terms: conditions — Infections; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Incidence of surgical site infection: The number of spinal surgery patients with surgical site infections.
  Interventions: Procedure: Spinal surgery

INTERVENTIONS:
Procedure: Spinal surgery — Elective spinal surgery performed

SUMMARY:
Post-operative wound infections can prolong hospital stays, increase rates of readmission to the intensive care unit, and increase the costs of treatment significantly. This study will conduct a prospective chart review of all patients undergoing elective spinal surgery on both the neurosurgery and orthopedic spine services at two facilities on an academic campus. The investigators will collect the data of those patients who develop post-surgical infections. This data will then be analyzed and compared to published data from other studies. The aim of this investigation is to passively collect this infection data, which may ultimately provide needed baseline incidence rates using current and standard protocols.

DETAILED DESCRIPTION:
This is a chart review study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing elective spinal surgery on either the neurosurgery and orthopedic spine services
* Patients who develop post-operative wound infections within 90 days of surgery

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients who are not undergoing elective spinal surgery on either the neurosurgery and orthopedic spine services
* Patients who do not develop post-operative wound infections within 90 days of surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older undergoing a spinal operation.
Sampling Method: Non-Probability Sample
Enrollment: 6959 (Actual)
Dates: Start 2011-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of patients who develop a surgical site infection (SSI) | 90 days following surgery
  Spinal reoperation at the same surgical location for incision, debridement and irrigation

CONTACTS AND LOCATIONS:
Overall Officials: Allan D Levi, MD, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No